CLINICAL TRIAL: NCT07037654
Title: Efficacy of Lingual Ondansetron in Reduction of Spinal Anesthesia-induced Hypotension In Cesarean Section; a Randomized Controlled Trial
Brief Title: Lingual Ondansetron in Reduction of Spinal Hypotension in Cesarean Section
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, professor of anaesthesia, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Lingual ondansetron
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hypotension After Spinal Anesthesia
Keywords: spinal anesthesia; lingual ondansetron; cesarean section

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ondansetron (Active Comparator): 8 mg of the lingual film form of ondansetron will be given 15 minutes before spinal anesthesia
  Interventions: Drug: ondansetron lingual film
- placebo (Placebo Comparator): a placebo lingual film form will be given 15 minutes before spinal anesthesia
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ondansetron lingual film — 8 mg of the lingual film form of ondansetron, given 15 minutes before spinal anesthesia
  Arms: ondansetron
Drug: Placebo — a placebo lingual film form, given 15 minutes before spinal anesthesia
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to learn if drug ondansetron, used in lingual form, lowers the incidence of spinal anesthesia-induced hypotension in cesarean sections. It will also learn about the safety of drug ondansetron. The main questions it aims to answer are

Does the drug ondansetron, used in lingual form, lower the incidence of spinal anesthesia-induced hypotension in cesarean sections? What medical problems do participants have when taking the drug ondansetron? Researchers will compare drug ondansetron to a placebo (a look-alike substance that contains no drug) to see if drug ondansetron works to reduce the incidence of spinal anesthesia-induced hypotension in cesarean sections

Participants will:

Take drug ondansetron or a placebo before induction of spinal anesthesia

DETAILED DESCRIPTION:
Spinal anesthesia, which is extensively used in a variety of surgical operations, frequently causes hypotension due to sympathetic nerve blocking. This reduction in blood pressure might have negative consequences, especially in people with cardiovascular comorbidities. Ondansetron, a selective serotonin 5-HT3 receptor antagonist, is well known for its antiemetic effects. However, its ability to reduce hypotension during spinal anesthesia has sparked great interest in recent years. Thus, it regulates cardiovascular function, vasodilation, and vascular tone and helps to maintain a more steady hemodynamic profile during spinal anesthesia.

A growing amount of evidence supports the use of ondansetron as a preventive strategy against spinal anesthesia-induced hypotension. This technique not only improves patient safety but also minimizes intraoperative problems. As research advances, using ondansetron in anesthetic protocols may become commonplace, reflecting its numerous benefits in the perioperative situation.

Objective: To investigate the efficacy of the lingual film form of ondansetron after use in parturients undergoing spinal anesthesia during cesarean delivery to reduce total ephedrine consumption and spinal-induced hypotension.

Methodology: Following the administrative ethical committee approval and informed patient consent obtained from 112 patients undergoing cesarean delivery in Suez Canal University Hospital, they will be randomly assigned to one of the two groups using a computer software program.

Group A (56 patients) will be administered 8 mg of the lingual film form of ondansetron, given 15 minutes before spinal anesthesia.

Group B (56 patients) will be administered a placebo lingual film form 15 minutes before spinal anesthesia.

Expected outcome: We can expect a reduction in the total ephedrine consumption and more cardiovascular stability based on the previous trial.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18- 40 years old parturients.
* Height: 150 to 180 cm
* Patients are ASA II (American Society of Anesthesiologists physical status grade II) = (pregnant and patients with mild systemic disease and no functional limitations).
* Patients scheduled for elective cesarean section in Suez Canal University Hospitals.

Exclusion Criteria:

* Patients' refused to participate in the study.
* Contraindications of spinal anesthesia (patients with marked deformities or infections at the site of spinal injection, and coagulopathy).
* Known allergy to bupivacaine or ondansetron.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only females undergoing ceserean sections
Enrollment: 112 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
ephidrine consumption | From the moment the surgery starts until it is finished, or after 90 minutes has passed, whichever is longer
  To evaluate the impact of lingual ondansetron on parturients having cesarean sections' overall intraoperative ephedrine consumption

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrhman Alshawadfy, Principal Investigator — Faculty of Medicine, Suez Canal University Ismailia, , Egypt
Locations (1):
- Faculty of Medicine, Suez Canal University, Ismailia, Egypt